CLINICAL TRIAL: NCT01278147
Title: Development and Implementation of a Cancer Fatigue Education Program
Brief Title: Cancer Fatigue Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de la Loire (Other)
Responsible Party: Professeur Franck Chauvin, Institut de Cancérologie de la Loire
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2007-A00147-46
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2011-01

CONDITIONS: Patient With Histologically Confirmed Malignancy
Keywords: cancer; fatigue program education
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- controle (No Intervention): patient without fatigue education program
- Education program (Experimental): the carer will help the patient develop competences on the following points: how to evaluate the severity of the fatigue; learn to recognize symptoms or prodromes showing associated difficulties (anxiety, fear, depression); how to improve control of fatigue by setting up suitable strategies (management of periods of activity and rest, physical and/or intellectual exercises, dietary program, complementary therapy); learn to ask for and accept the help of close relations or carers.
  Interventions: Behavioral: fatigue education program

INTERVENTIONS:
Behavioral: fatigue education program — the carer will help the patient develop competences on the following points: how to evaluate the severity of the fatigue; learn to recognize symptoms or prodromes showing associated difficulties (anxiety, fear, depression); how to improve control of fatigue by setting up suitable strategies (management of periods of activity and rest, physical and/or intellectual exercises, dietary program, complementary therapy); learn to ask for and accept the help of close relations or carers.
  Arms: Education program

SUMMARY:
The purpose of the present project is to develop, implement and evaluate a pilot regional patient education program on the management of one of the main side effects of chemotherapy in cancer patients, that is fatigue.

A carer (doctor or nurse) trained in educational techniques will be responsible for the patient. The carer will first identify modes of behavior and competences that the patient must acquire in order to optimize his/her management of fatigue ("educational diagnosis"). An education program, based on a contract of goals will be proposed after this diagnosis phase. The expected results are, in the short-term, a significant reduction in the mean level of fatigue in patients receiving chemotherapy who benefited from individual educational management. In the longer term, the aim is to evaluate the impact of this program on patient quality of life and use of healthcare structures in comparison with conventional management.

ELIGIBILITY:
Inclusion Criteria:

* - Age> 18 years.
* Patient with histologically confirmed malignancy, during initial treatment with chemotherapy, followed or not by surgery, or the first week of radiotherapy. Patients with hematologic malignancy (including non-Hodgkin's lymphoma or Hodgkin's disease) may be included in the study, except for patients with leukemia.
* Having a fatigue up during the week preceding the inclusion level measured by the average patient with 2 or more on a visual analogue scale (VAS) graded from 0 to 10 (0 expressing no fatigue and 10 the maximum fatigue imaginable ).
* Volunteered to participate in PEPs "Coping with fatigue."
* Usually followed as outpatients.
* Condition preserved (ECOG PS 2).
* Available for all meetings of the educational program (5 sessions of 2 hours over a period of 5 weeks).
* Able to read, write and understand French.
* Resident (s) in a 50 km radius around the center investigator.
* Can be contacted by phone.
* Compulsory membership of a social security system.
* Obtaining informed consent in writing, signed and dated.

Exclusion Criteria:

* - Patient (e) with the inclusion anemia with a hemoglobin level below 10 g/100 mL.
* Patient (e) having a documented history of cognitive or psychiatric disorders.
* Patient (e) can not be followed for family, social, geographical or psychological.
* Patient (e) deprived of their liberty by court or administrative

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2007-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Education program | 8 weeks
  The main indicator of patient satisfaction after the education program will be the change during 8 weeks of follow-up in the mean fatigue score measured on a specific scale (FACT-F) (32).

SECONDARY OUTCOMES:
self-evaluation | 8 weeks
  One secondary efficacy variables will comprise self-evaluation of patient quality of life measured using the SF-36 scale
healthcare structures | 8 weeks
  The secondary efficacy variables will comprise evaluation of the use by patients of healthcare structures (phone calls, number of home visits, number of days of hospitalization, visits to emergency departments, other carers).

CONTACTS AND LOCATIONS:
Overall Officials: Franck CHAUVIN, Pr, Principal Investigator — Institut de Cancérologie de la Loire
Locations (7):
- France (7):
  - PIVOT, Besançon
  - CHOLLET, Clermont-Ferrand
  - ZANETTA, Dijon
  - BACHELOT Thomas, Lyon
  - BLAY, Lyon
  - LAFONT, Lyon
  - CLAVREUL, Saint-Etienne